CLINICAL TRIAL: NCT00528450
Title: Phase II Study of Combined All-Trans Retinoic Acid and Arsenic Trioxide for Acute Promyelocytic Leukemia Followed by Risk-Adapted Postremission Therapy
Brief Title: Tretinoin and Arsenic Trioxide With or Without Idarubicin in Treating Patients With Acute Promyelocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-108; P30CA008748 (NIH); MSKCC-07108; CEPHALONO-MSKCC-07108
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Leukemia
Keywords: adult acute promyelocytic leukemia (M3); adult acute myeloid leukemia with t(15;17)(q22;q12); untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide; Idarubicin; Tretinoin

ARMS (1):
- Tretinoin and Arsenic Trioxide With or Without Idarubicin (Experimental): See Outline for details
  Interventions: Drug: arsenic trioxide; Drug: idarubicin; Drug: tretinoin

INTERVENTIONS:
Drug: arsenic trioxide
Drug: idarubicin
Drug: tretinoin

SUMMARY:
RATIONALE: Tretinoin may help cancer cells become more like normal cells, and to grow and spread more slowly. Drugs used in chemotherapy, such as arsenic trioxide and idarubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving tretinoin together with arsenic trioxide with or without idarubicin may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving tretinoin together with arsenic trioxide with or without idarubicin works in treating patients with acute promyelocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the rate of molecular remission after induction therapy comprising tretinoin (ATRA) and arsenic trioxide (ATO) (along with idarubicin in patients with leukocytosis) in patients with acute promyelocytic leukemia (APL).

Secondary

* To determine the rate of clinical complete remission and the time to remission after induction therapy.
* To determine the proportion of patients in molecular remission after each course of postremission therapy and to use these findings to direct the number of consolidation courses with ATRA and idarubicin that are administered.
* To determine the disease-free survival and overall survival of patients treated with this regimen.
* To determine the toxicity of this treatment regimen, including the number and length of hospitalizations, the incidence of secondary myelodysplastic syndromes or acute myeloid leukemia, and the effects of treatment on LVEF.
* To characterize the differentiation of APL cells during treatment with combined ATRA and ATO using serial immunophenotyping studies of peripheral blood and bone marrow.
* To compare the results of quantitative real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assays performed on bone marrow and peripheral blood.

OUTLINE:

* Induction therapy: Patients receive tretinoin orally twice daily and arsenic trioxide IV over 1-4 hours once daily until a marrow remission is documented or for 60 days, whichever comes first. Patients with leukocytosis (WBC > 10,000/μL) also receive idarubicin IV over 10-15 minutes beginning on day 2 and continuing every other day for 4 doses. Patients who achieve a clinical complete remission (CR) proceed to consolidation therapy. If a marrow remission is not achieved after 60 days, the patient is removed from the study.
* Consolidation therapy:

  * Consolidation courses 1, 2, and 3: Beginning 3-6 weeks after documentation of clinical CR, patients receive consolidation therapy comprising tretinoin orally twice daily for 15 days and arsenic trioxide IV over 1-4 hours once daily 5 days a week for 5 weeks. Consolidation therapy repeats every 3-6 weeks for 3 courses.

Patients who have a negative PML-RARα transcript by reverse transcriptase-polymerase chain reaction (RT-PCR) assay after consolidation course 2 proceed to maintenance therapy after receiving consolidation course 3. Patients who have a negative PML-RARα transcript by RT-PCR assay after consolidation course 3, proceed to consolidation course 4 followed by maintenance therapy. Patients who have a positive PML-RARα transcript by RT-PCR assay after consolidation courses 2 and 3 proceed to consolidation courses 4 and 5.

* Consolidation course 4: Beginning 3-6 weeks after completion of consolidation course 3, patients receive tretinoin orally twice daily for 15 days and idarubicin IV over 10-15 minutes once daily for 4 days.
* Consolidation course 5: Beginning 3-6 weeks after completion of consolidation course 4, patients receive tretinoin orally twice daily for 15 days and idarubicin IV over 10-15 minutes once daily for 3 days.

Patients who remain positive for the PML-RARα transcript after 5 courses of consolidation therapy are removed from the study. Patients who have a negative PML-RARα transcript after 5 courses of consolidation therapy proceed to maintenance therapy.

* Maintenance therapy: Beginning approximately 3 months after completion of the final consolidation course, patients receive tretinoin orally twice daily for 15 days. Treatment repeats every 3 months for up to 2 years.

Disease status will be monitored with serial analyses of bone marrow and peripheral blood samples using RT-PCR for PML-RARα mRNA. Patients will be followed until relapse, death, loss to follow-up, or removal from study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologic diagnosis of acute promyelocytic leukemia (APL), confirmed by one of the following:

  * Demonstration of t(15;17) using conventional cytogenetics or fluorescence in situ hybridization (FISH)
  * Positive PML-RARα transcript by reverse transcriptase-polymerase chain reaction (RT-PCR) assay
* Patients with CNS involvement by APL are eligible

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Creatinine ≤ 2.0 mg/dL or creatinine clearance > 60 mL/min
* Bilirubin < 2.0 mg/dL (unless attributed to Gilbert disease)
* Alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN)
* AST and ALT ≤ 2.5 ULN
* LVEF ≥ 50% on echocardiogram or MUGA scan
* QTc ≤ 500 msec on baseline ECG
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 4 months after the completion of study treatment
* No active serious infections not controlled by antibiotics
* No other concurrent active malignancy requiring immediate therapy
* No clinically significant cardiac disease (New York Heart Association class III or IV heart disease), including chronic arrhythmias
* No pulmonary disease
* No other serious or life-threatening condition deemed unacceptable by the principal investigator

PRIOR CONCURRENT THERAPY:

* No prior treatment for APL

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G. Jurcic, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Peter Maslak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Tretinoin and Arsenic Trioxide With or Without Idarubicin
Period: Overall Study
Arm/Group | All Patients
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Molecular Remission Rate
Description: # of patients with Complete Remission
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=1)
ALT, SGPT (Blood and lymphatic system disorders) | 1 (1)
AST, SGOT (Blood and lymphatic system disorders) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Infection, other (Infections and infestations) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Mood alteration - Anxiety (Psychiatric disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Pain - Head/headache (General disorders) | 1 (1)
Pain - Pain NOS (General disorders) | 1 (1)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes